CLINICAL TRIAL: NCT06963983
Title: Personalized Rehabilitation System Using Gamification With Virtual Reality Technology: A Feasibility Study
Brief Title: Virtual Reality Rehabilitation for Shoulder Pathologies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Dr. Alexandre Lädermann, Orthopaedic surgeon, La Tour Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00166
Record Dates: First submitted 2025-04-23; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Shoulder Instability; Frozen Shoulder; Rotator Cuff Tears
MeSH Terms: conditions — Bursitis; Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Shoulder Pathology Group (Experimental): Patients suffering from either shoulder instability, frozen shoulder or rotator cuff tears
  Interventions: Device: Rehabilitation using virtual reality

INTERVENTIONS:
Device: Rehabilitation using virtual reality — During the four physiotherapy (PT) sessions (60 min for each session), a set of exercises from the conventional PT is replaced by multiple short sessions of 30 minutes each, where the patient will be equipped by a set of motion trackers mounted on a belt and on a set of straps to be worn around both arms and both forearms. The patient will also hold a controller in each hand and wear a commercial VR headset on his head. Then, thanks to the headset, the patient will be able to experience a set of VR environments, where he or she will be guided through a set of exergames. His/her movements in the real world will be used to move his/her avatar's body in the virtual world, and the exergames will be designed to push him/her to perform the motions required by the therapy in order to go through the games. Various strategies, including a virtual coach will also appear to prevent the patient from doing potentially hazardous movements.

SUMMARY:
Most rehabilitation protocols require patients to train the affected limbs with high regularity, following repetitive cycles of exercises, in order to recover mobility and strength. Nonetheless, the repetitive nature of these exercises can demotivate patients leading to less intense and committed training, if not ending with a lack of compliance toward the prescribed exercises, ultimately leading to a suboptimal recovery. For this reason, several research groups are investigating solutions to help patients in this process, using robotic support or protocols assisted by virtual reality (VR).

Most of these studies have shown benefits, notably in the field of post-stroke rehabilitation, however numerous types of physical therapies have not been investigated yet. Therefore, the main goal of this study will be to explore if the combination of modern motion-tracking and VR can provide significant functional outcomes for the treatment of the most common upper limb pathologies. The investigators created a set of exergames designed to lead the patients through a gamified version of part of physiotherapy (PT). This modified therapy is expected to offer several benefits to the treatment with respect to a purely conventional therapy: (i) improved patient's motivation and commitment to the exercises; (ii) constant evaluation of the patient's performance, thanks to the use of motion tracking; (iii) session-by-session tuning of exercises difficulty; (iv) clear progress traceability; (v) real-time alerts in case of problematic or compensatory movements; (vi) measurement and evaluation of new metrics of movements quality that were not possible in conventional therapy setups.

To evaluate the feasibility of this project, the investigators would like to test the VR system on a short series of patients during four sessions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients able to understand the content of the patient information / consent form and give consent to take part in the research project
* Glenohumeral instability surgical treated with traumatic initial instability in a < 20 years old athlete, recurrent instability with one or more of the following criteria: a failure of conservative treatment, locked dislocation, failed prior surgery, high risk for further recurrence (i.e. collision or competitive athletes), Critical glenoid bone-loss (>15-20%), bipolar bone-loss resulting in "off-track" lesion
* Partial or complete rotator cuff repair with an indication to postoperative rehabilitation depending on surgeon recommendation
* Idiopathic, primary, or secondary frozen shoulder

Exclusion Criteria:

* Patients with a language barrier hindering questionnaires completion
* Patients unlikely to attend clinical follow-up (e.g. when living abroad)
* Legal incompetence
* Enrolment of the investigators, his/her family members, employees and other dependent persons
* Non-motivated patients
* Active infection
* Exclusion criteria related to glenohumeral instability: uncontrolled epilepsy, spontaneous unidirectional instability in a hyperlax patient, multidirectional instability, elher-Danlos syndrome
* Exclusion criteria related to rotator cuff tears: Additional procedure(s) (muscle transfer, patch,…)
* Exclusion criteria related to VR use: Patients with a predisposition to motion sickness, Patients suffering from epilepsy or having any serious mental illness (schyzophrenia, neurological problems, etc.), Patients with visual impairment , Patients will intellectual disability that prevent them to understand how to use the VR rehabilitation system, Patients with bilateral upper limb injuries, as one side is needed as healthy reference

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Simulator Sickness Questionnaire | Day 1
  From 1 (best) to 7 (worst)

SECONDARY OUTCOMES:
A reduced version of the Post-experimental Intrinsic Motivation Inventory | Day 1
  From 1 (worst) to 7 (best)
A reduced version of the Avatar Embodiment Questionnaire | Day 1
  From 1 (worst) to 7 (best)
Patient satisfaction | Day 1
  4-Point Likert Scale (Not satisfied at all, Not satisfied, Satisfied, Very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lädermann, MD, Principal Investigator — La Tour hospital, Meyrin (1217) Geneva, Switzerland
Locations (1):
- La Tour hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No